CLINICAL TRIAL: NCT07172568
Title: Randomisierte, Kontrollierte Untersuchung Der Wirksamkeit Von Blood Flow Restriction (BFR)-Training Zur Behandlung Der Epicondylopathia Humeri Radialis
Brief Title: Blood Flow Restriction Training For The Treatment Of Lateral Epicondylopathy
Acronym: EPIC-BFR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 245/21 S-NP
Record Dates: First submitted 2023-02-13; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Elbow Tendinopathy; Elbow, Tennis; Lateral Epicondylitis; Epicondylitis of the Elbow; Blood Flow Restriction Therapy; BFR
Keywords: Randomised controlled Trial; RCT; Interventional study; BFR; Blood-Flow-Restriction-Therapy; lateral Epicondylopathy; Epicondylitis
MeSH Terms: conditions — Elbow Tendinopathy; Tennis Elbow | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: It's a Randomized Controlled Trial, double blinded. The participant and the investigator are blinded and have no information about the group affiliation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The Participant is randomly assigned to a cohort by drawing a number. Only the attending physiotherapist knows which number belongs to which cohort and start then either the BFR-training or the sham-BFR. The examining doctor in the preliminary investigation and in the follow-ups does not know how the patients were treated. Also the outcomes assessor has no informations about the treatment of the patients, therefore the assessment of the results is also carried out blindly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 20mmHg pressure Blood Flow Restriction (Active Comparator): The patients in the control group are wearing a blood-flow-restriction cuff proximal to the elbow with an applied pressure of just 20mmHg. Studies have shown that this amount of pressure has no impact. The control group remains blind using the cuff with low pressure. The therapy protocol is exactly the same as in the Interventional group.
  Interventions: Procedure: sham-Blood Flow Restriction
- 50% of Mean arterial blood pressure Blood Flow Restriction (Experimental): The patients in the intervention group are wearing a blood-flow-restriction cuff proximal to the elbow with an applied pressure of 50% of the mean arterial blood pressure. The therapy protocol is exactly the same as in the control group.
  Interventions: Procedure: Blood Flow Restriction

INTERVENTIONS:
Procedure: Blood Flow Restriction — In the intervention group, 50% of limb occlussion pressure are applied to the extremity during exercises.
  Arms: 50% of Mean arterial blood pressure Blood Flow Restriction
Procedure: sham-Blood Flow Restriction — In the control group, 20 mmHg are applied to the extremity during exercises.
  Arms: 20mmHg pressure Blood Flow Restriction

SUMMARY:
The study aims to evaluate the effectiveness of Blood Flow Restriction Training for the treatment of lateral elbow epicondylopathy.

DETAILED DESCRIPTION:
1. To test a non-invasive, rapid treatment option for epicondylopathia humeri radialis for its effectiveness, Blood Flow Restriction (BFR) training will be supplemented to the applied exercise therapy. In BFR training, blood flow to the muscle is reduced by tying off the limb to be trained, e.g. with a blood pressure cuff, to achieve mechanical compression of the underlying blood vessels. This results in increased accumulation of blood in the capillary bed distal to the pressure cuff. Although isolated adverse effects have been reported, based on the current literature, it can be assumed that BFR training is comparable to conventional training in terms of safety for the user. Regarding the effect of BFR applications, it has been shown that even BFR without additional training measures can reduce muscle atrophy occurring during immobilization. A systematic literature review confirmed the positive effect of BFR augmented strength training in terms of strength development as well as muscle gain. The first positive results of BFR training compared to conventional physiotherapy have already been shown in rehabilitation after replacement surgery of the anterior cruciate ligament and after treatment of a radius fracture. Therefore, there is a scientific interest to verify the effectivity of this method in another disease of the musculoskeletal system, epicondylopathia humeri radialis.

   Question: Does the implementation of a BFR-protocol in the physiotherapeutic treatment of epicondylopathia humeri radialis lead to a significantly pain relief and function improvement in the affected hand? Hypothesis: The implementation of a BFR-protocol in the physiotherapeutic treatment leads to a significantly pain relief an function improvement in comparison to a cohort without BFR.
2. All patients who meet the inclusion criteria will be informed about the study in the special consultation for shoulder and elbow diseases and asked whether they would like to participate and will receive a declaration of participation if they agree. Patients are informed in detail that participation is voluntary, and that non-participation will not result in any disadvantages for their treatment. Prior to the start of therapy, one of the above-mentioned study physicians will personally inform the patient about the risks and benefits of the study. After sufficient time for reflection, the corresponding declaration of participation is gone through with the patient, signed by both parties in case of consent and the patient receives a copy of it. After signing the participation form, an appointment will be made to start the six-week randomized physiotherapy (2x per week a 20min; group A: Physiotherapy + BFR while intermittently wearing the BFR cuff (Delfi Medical Innocation Inc., Vancouver, Canada) at 50% of arterial occlusion pressure analogous to previous studies; Group B Physiotherapy + sham-BFR (BFR cuff inflated to 20mmHg). Patients are informed that they can discontinue therapy without giving a reason.

Physiotherapy treatment will be performed according to the current evidence-based protocol in the Department and Polyclinic for Sports Orthopedics of the Klinikum rechts der Isar of the Technical University of Munich twice a week over a period of six weeks. Randomization will be done by the treating physiotherapist(s) before the first physiotherapy session. Before the start of the first therapy unit (T1), as well as after completion of the six-week intervention (T2), six weeks after completion of therapy (T3) and again 12 weeks aufter completion of the physiotherapeutic treatment (T4), both clinical examinations to assess the progress of therapy by a blinded study physician and the completion of a standardized questionnaire by the subject will take place. No travel or expense allowance is provided. During the clinical examination, the joint status as well as the clinical signs of epicondylopathia radialis humeri will be collected. Further data collection is performed by means of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of lateral epicondylitis
* duration of symptoms > 6 weeks
* failed physical therapy
* absence of x-ray abnormalities
* written and informed consent

Exclusion Criteria:

* prior joint infiltrations
* duration of symptoms > 12 months
* concomitant rheumatoid diseases
* concomitant elbow pathologies, including medial epicondylitis
* concomitant radicular symptoms of the cervical spine, shoulder or hand
* traumatic etiology of symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale for pain | 3 months
  VAS at rest and at dorsal extension of the hand. Measuring the pain on a scale from 1-10. 1 means no pain and 10 means extreme pain. The investigators are measuring the pain on the VAS scale once before and three times after the intervention within a time frame of 3 Months (directly after the intervention, 6 weeks after the intervention and 12 Weeks after the intervention).
  A higher score means a worse outcome, a lower score means a better outcome.
Mayo Elbow Performance Score | 3 Months
  The Mayo Elbow Performance Score (MEPS) is a clinical tool used to assess the function of the elbow joint, particularly in patients with elbow disorders or after treatment (e.g., surgery). It evaluates pain, range of motion, function, and elbow stability.
  Range of Scores: 0 to 100. 100 represents excellent elbow function with no pain. 75-89 is considered good, 60-74 is fair, and below 60 is poor.
  Scores are assessed before and three times after the intervention:
  Immediately post-intervention. 6 weeks post-intervention. 12 weeks post-intervention. This allows tracking of elbow recovery and functional improvement over time. A higher score indicates better recovery and elbow function.
Short-form 36 questionnaire (SF-36) | 3 Months
  It is a questionnaire which is answered by the patients. The SF-36 (Short Form 36) Health Survey is a widely used questionnaire designed to assess an individual's overall health status. It measures eight domains of health:
  Physical Functioning Role Physical Role Emotional Mental Health Vitality (Energy/Fatigue) Social Functioning Pain General Health Each domain is scored on a scale from 0 to 100, with 0 representing the worst health status and 100 representing the best. The scores are then used to evaluate physical and mental health, as well as the impact of health on daily functioning.
  Range of Scores: 0-100 for each domain. Higher scores represent better health and functioning. Lower scores indicate greater impairment or worse health status. It helps in understanding an individual's quality of life and the impact of disease or disability on their physical and mental well-being.
  It is commonly used to evaluate patient health outcomes.
Disabilities of the Arm, Shoulder and Hand questionnaire | 3 Months
  The DASH (Disabilities of the Arm, Shoulder, and Hand) questionnaire is a tool used to assess the physical function and symptoms in patients with musculoskeletal disorders of the upper limb. It evaluates function and pain in daily activities.
  Range of Scores: 0 to 100. 0 represents no disability (full function, no pain). 100 represents maximum disability (severe limitation and pain).
  The DASH score is typically measured before and three times after an intervention:
  Immediately post-intervention. 6 weeks post-intervention. 12 weeks post-intervention. Lower scores indicate better function and less disability, while higher scores show greater functional impairment and pain. The DASH helps to monitor recovery and the effectiveness of treatments for upper limb conditions.
Patient rated tennis elbow evaluation questionnaire | 3 Months
  The Patient-Rated Tennis Elbow Evaluation (PRTEE) is a questionnaire specifically designed to assess the severity of symptoms and the impact of lateral epicondylitis (tennis elbow) on a patient's daily life. It evaluates pain and function in the elbow, particularly in activities related to gripping and arm movement.
  Range of Scores: 0 to 100. 0 represents no pain or disability. 100 represents maximum pain or disability.
  The PRTEE is typically assessed before and three times after an intervention:
  Immediately post-intervention. 6 weeks post-intervention. 12 weeks post-intervention. Lower scores indicate less pain and disability, while higher scores suggest greater severity of symptoms. It is used to track the patient's progress and recovery from tennis elbow over time.
clinical evaluation of the elbow | 3 Months
  clinical Evaluation including: Range of Motion
Strength-Measurement: Dorsal extension of the hand | 3 Months
  Strength-Measurement: Dorsal extension of the hand using a dynamometer (MicroFET 2, Hoggan Scientific, Salt Lake City, USA). Measuring the affected elbow and the non-affected elbow
Drop-Out | 3 Months
  statistical measurement of patients drop-out-quote using a Questionnaire about potential change to surgical Interventions or another type of therapy.
  statistical measurement of Lost to follow-up patients
clinical examination of the elbow | 3 Months
  A clinical examination of the elbow is performed. The focus here is on the examination of possible instability in the elbow joint. To this end, valgus-axis stress is applied and the ability to open the joint is checked.
  The examination is assessed before and three times after an intervention:
  Foldability and instability indicate a poor outcome
clinical evaluation of the elbow | 3 Months
  clinical evaluation of the elbow using Epicondylitis Tests (Cozen-Test)
clinical evaluation of the elbow | 3 Months
  clinical evaluation of the elbow using Epicondylitis Tests (Reversed-Cozen-Test)
clinical evaluation of the elbow | 3 Months
  clinical evaluation of the elbow using Epicondylitis Tests (Maudsley-Test)
clinical examination of the elbow | 3 Months
  A clinical examination of the elbow is performed. The focus here is on the examination of possible instability in the elbow joint. To this end the milking maneuver is examined with possible medial opening.
  The examination is assessed before and three times after an intervention:
  Foldability and instability indicate a poor outcome
clinical examination of the elbow | 3 Months
  A clinical examination of the elbow is performed. The focus here is on the examination of possible instability in the elbow joint. To this end the tweezer grip on the elbow are examined.
  The examination is assessed before and three times after an intervention:
  Foldability and instability indicate a poor outcome
clinical examination of the elbow | 3 Months
  A clinical examination of the elbow is performed. The focus here is on the examination of possible instability in the elbow joint. To this end the pivot-shift test on the elbow is examined.
  The examination is assessed before and three times after an intervention:
  Foldability and instability indicate a poor outcome
clinical examination of the elbow | 3 months
  A clinical examination of the elbow is performed. The focus here is on the examination of possible instability in the elbow joint. To this end, varus-axis stress is applied and the ability to open the joint is checked.
  The examination is assessed before and three times after an intervention:
  Foldability and instability indicate a poor outcome

SECONDARY OUTCOMES:
Questionnaire | 3 Months
  The questionnaire the investigators created, also contains individual questions that ask about possible confounders. These are questions about gender
  * Age
  * Nicotine abuse
  * Type of sport, activity level/intensity, frequency with these questions the investigators would like to identify possible confounders.
Body mass index (BMI) | 3 Months
  measuring secondary objective as a potential confounder
Return-to-sports | 3 Months
  The Return to Sports Rate is a measure used to assess the percentage of individuals who return to their pre-injury or pre-intervention level of sports activity following treatment or rehabilitation. It provides insight into how effectively a patient has recovered and whether they can resume their sports participation at a similar level to before the injury.
  In this case, the investigators use a questionnaire to gather information about the type of sport, frequency, and weekly time commitment to sports activities.
  By comparing the responses from these time points, the investigators can calculate the Return to Sports Rate. This rate is determined by assessing how many participants have returned to their previous levels of sports activity, or how close they are to their baseline sports participation after the intervention.
Return-to-work | 3 Months
  The Return to Work Rate is a measure used to assess the percentage of individuals who are able to return to their pre-injury or pre-intervention work activities following treatment or rehabilitation. It helps to evaluate the effectiveness of the intervention in enabling patients to resume their work duties. In this case, the investigators use a questionnaire to gather information about the type of work, work frequency, and the time commitment per week spent on work activities.
  By comparing the responses from these time points, the investigators can calculate the Return to Work Rate. This rate is determined by assessing how many participants have returned to their previous work activities or how close they are to their baseline work participation after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Hinz, MD, Principal Investigator — Department of Sports Orthopaedics, Technical University of Munich
Locations (1):
- Department of Sports Orthopaedics, Technical University of Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
IPD is not shared due to strict data protection laws in Germany, such as the GDPR, which ensure the security of sensitive medical data. Sharing individual patient data poses significant risks to data security, particularly regarding unauthorized access or misuse. Additionally, explicit consent from participants is often missing for data sharing beyond the original research purpose. Without such consent, any disclosure would be legally impermissible and ethically problematic. Therefore, safeguarding privacy and complying with legal regulations are paramount.

REFERENCES:
- [Background] Hinz M, Franz A, Pirker C, Traimer S, Lappen S, Doucas A, Siebenlist S. [Blood flow restriction training as a treatment option for lateral elbow tendinopathy-a study presentation]. Orthopadie (Heidelb). 2023 May;52(5):365-370. doi: 10.1007/s00132-023-04370-w. Epub 2023 Apr 20. German. PMID 37079041
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37079041/